CLINICAL TRIAL: NCT03820141
Title: Multicenter Phase II Trial of Durvalumab (MEDI4736) with Trastuzumab and Pertuzumab Combination in HER2-Enriched and HER2-Amplified Breast Cancer (DTP Trial)
Brief Title: Durvalumab with Trastuzumab and Pertuzumab in HER2-Enriched Breast Cancer
Acronym: DTP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Polly A. Niravath, MD, Oncologist, Houston Methodist Neal Cancer Center, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00020917
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab + Trastuzumab + Pertuzumab (Experimental): Durvalumab, trastuzumab, and pertuzumab will be administered on Day 1 every 3 weeks for 6 cycles. Trastuzumab will be administered as 8 mg/kg intravenous (IV) loading dose, followed by 6 mg/kg IV. Pertuzumab will be administered as 840 mg IV loading dose, followed by 420 mg. Durvalumab will be administered at a fixed dose of 1120 mg IV.
  Interventions: Drug: Durvalumab; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Durvalumab — programmed cell death-ligand 1 inhibitor
  Other Names: IMFINZI, MEDI4736
Drug: Trastuzumab — anti-HER2 monoclonal antibody
  Other Names: Herceptin
Drug: Pertuzumab — anti-HER2 monoclonal antibody
  Other Names: Perjeta

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of using durvalumab with trastuzumab and pertuzumab in participants with human epidermal growth factor receptor 2 (HER2)-enriched breast cancer.

DETAILED DESCRIPTION:
The purpose of this research study is to test the safety and effectiveness of using durvalumab with trastuzumab and pertuzumab in participants with HER2-enriched breast cancer. The standard or usual pre-surgery treatment for this type of disease are drugs called trastuzumab and pertuzumab that target HER2. Studies have shown that trastuzumab and pertuzumab treatment can stimulate the body's own immune system to attack cancer cells. Durvalumab is a drug that also activates the immune system. The use of durvalumab together with trastuzumab and pertuzumab treatment may allow the immune system to work harder to kill cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged >18 years at the time of study entry.
2. Histologically confirmed HER2-enriched (by BluePrint) and HER2-amplified (ERBB2 mRNA >7.5-10) breast cancer.
3. Estrogen receptor and progesterone receptor negative.
4. Primary tumor greater than 1 cm diameter, measured by clinical examination and mammography or echography.
5. Any nodal status
6. Bilateral breast cancers that individually meet eligibility criteria are allowed.
7. Eastern Cooperative Oncology Group performance status of 0 or 1.
8. Adequate organ and marrow function.
9. Baseline left ventricular ejection fraction greater than or equal to 50%, as measured by multigated acquisition scan or echocardiogram.
10. Evidence of postmenopausal status or negative serum pregnancy test for premenopausal patients. Negative serum beta-human chorionic gonadotropin pregnancy test within 7 days prior to the first dose of study treatment for premenopausal patients.
11. Willing to provide biopsy tissues as required by the study.
12. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product within 28 days prior to the first dose of study treatment.
2. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
3. Unresolved or unstable adverse events from prior administration of another investigational drug.
4. Any concurrent chemotherapy, radiation therapy, immunotherapy, or biologic therapy for cancer treatment.
5. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of study treatment.
6. History of allogenic organ transplantation.
7. Active or prior documented autoimmune or inflammatory disorders.
8. History of active primary immunodeficiency.
9. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.
10. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study treatment.
11. Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment.
12. Patients who are pregnant or breastfeeding or patients of reproductive potential who are not willing to employ effective birth control from screening to 7 months after the last dose of study treatment.
13. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
14. Patients with a mean QT interval of greater than or equal to 470ms calculated from 3 EKGs
15. Patients with underlying cardiovascular conditions that have recently undergone interventions including: cardiac ventricular arrhythmia requiring medication, history of second or third degree AV blocks, myocardial infarction with the previous year, congestive heart failure, and unstable angina
16. Patients with a LVEF less than 50%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate in the breast in patients with HER2-enriched and HER2-amplified breast cancer | 18 weeks
  Determine pCR rate in the breast in patients with HER2-enriched and HER2-amplified breast cancer

SECONDARY OUTCOMES:
pCR rate in the breast in patients whose tumors have <5% and ≥5% tumor-infiltrating lymphocytes (TILs) | 18 weeks
  Determine pCR rate in the breast in patients whose tumors have <5% and ≥5% TILs
pCR rate in patients with programmed cell death-ligand 1 (PD-L1)-positive and PD-L1-negative tumors | 18 weeks
  Determine pCR rate in the breast in patients with PD-L1-positive and PD-L1-negative tumors
Three-year disease-free survival (DFS) rate in patients who achieve pCR | 3 years
  Determination of 3-year DFS rate in patients who achieve pCR
Number of participants with treatment-related adverse events | 18 weeks
  Number of participants with treatment-related adverse events, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Polly Niravath, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No